CLINICAL TRIAL: NCT01960231
Title: The Effect of ß-cell Specific Glucokinase Mutation on Glucose Homeostasis and Insulin Secretion in a MODY-2 Family
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Sponsor
Other Study IDs: SHEBA-13-0464-JI-CTIL
Record Dates: First submitted 2013-09-30; First posted 2013-10-10 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: MODY-2 Diabetes
MeSH Terms: interventions — Glucose Tolerance Test

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- pancreas specific MODY-2
  Interventions: Other: OGTT

INTERVENTIONS:
Other: OGTT

SUMMARY:
Type 2 diabetes mellitus patients exhibit many glucose homeostasis abnormalities in different tissues and organs. Among the more important defects are disturbed hepatic glucose metabolism and defective pancreatic β-cell function. Hexokinase IV, commonly known as glucokinase, is the predominant hexokinase expressed in the liver, the pancreatic β-cells (where it functions as the glucose sensor for insulin secretion) and in glucose-sensory cells in the hypothalamus and gut.

The glucokinase gene contains two distinct promoters. The downstream one is active only in hepatocytes and the upstream promoter is active only in extrahepatic glucose sensory-cells. Alternative promoters enable differential regulation of gene transcription in liver and extrahepatic sites. In pancreatic β-cells, glucokinase expression at the mRNA level is largely constitutive, whereas in the liver it undergoes large adaptive changes in response to nutritional states, enabling larger changes in glucokinase activity than would otherwise be possible by post-transcriptional regulation alone.

Most of the MODY-2 patients were found to have glucokinase mutations located in areas that are common to the liver and pancreas. The diabetes in these patients is related both to defect in insulin secretion and abnormal hepatic glucose metabolism. Point mutation in the pancreatic specific promoter was recently described as a cause for impaired fasting glucose [Diabetes 58:1929-1935, 2009]. The investigator have recently identified a MODY-2 family with a genetic defect that is located in the pancreatic promoter, sparing the liver promoter. This family demonstrates that abnormal insulin secretion alone (perhaps together with other extrahepatic glucose sensors) is enough to cause diabetes.

In this study, the investigators would like to use an oral glucose tolerance test (OGTT) and continuous glucose monitoring (CGM) technique in order to elucidate the relative roll of the hepatic glucokinase in normal glucose homeostasis. This issue is complicated by the fact that in addition to glucokinase, hexokinase isoenzymes I, II and III are also expressed at very low levels in hepatocytes. They are an important back-up mechanism when glucokinase activity is compromised, as in liver cirrhosis or murine models with liver-specific glucokinase knock-down. However, impaired hepatic glycogen synthesis was demonstrated in MODY-2 subjects (JCI 1996:98:1755). By comparing members of the investigators MODY-2 family with members of other MODY-2 families and normal controls the investigators hope to shade some light on this question.

ELIGIBILITY:
Inclusion Criteria:

1. MODY 2 patients with documented mutations in the glucokinase promoter or coding region.
2. Healthy non-diabetic individuals matched for age, sex and BMI with recruited MODY2 patients.
3. Age range - 12-80; males and females

Exclusion Criteria:

1. Unable to provide written informed consent.
2. Unable to safely stop glycemia related medications for the duration of the test + wash-out period.

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: MODY-2 family
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
fasting and post glucose load glucose level | 1 year

SECONDARY OUTCOMES:
fasting and post glucose load Insulin | 1 year
fasting and post glucose load c-peptide | 1 year

OTHER OUTCOMES:
glucose metabolism measured by CGMS | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Ilany, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Ramat Gan, Israel